CLINICAL TRIAL: NCT00592852
Title: A Pilot Treatment Study of Fluoxetine for Obsessive-Compulsive Disorder in Children and Adolescents With Bipolar Disorder
Brief Title: Fluoxetine for Obsessive-Compulsive Disorder in Children and Adolescents With Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow subject recruitment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Clinical Investigator, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-P-001840
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2012-03-06 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Bipolar Disorder; Pediatric OCD
Keywords: bipolar disorder; obsessive compulsive disorder; Prozac
MeSH Terms: conditions — Bipolar Disorder; Obsessive-Compulsive Disorder | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoxetine (Experimental)
  Interventions: Drug: fluoxetine

INTERVENTIONS:
Drug: fluoxetine — capsules, dose range of 10mgQD - 60mgQD, given daily for 12 weeks
  Other Names: Prozac

SUMMARY:
This will be a 12-week open-label pilot treatment study for children and adolescents (ages 6-17) who meet DSM-IV criteria for bipolar disorder (BPD) and obsessive-compulsive disorder (OCD) who are adequately mood stabilized on a stable regimen based on standard clinical care. Specific hypotheses are as follows:

Hypothesis 1: Children and adolescents with comorbid OCD and BPD who have achieved adequate mood stabilization using a naturalistic clinical practice approach, will benefit from an FDA-approved selective seratonin reuptake inhibitor (SSRI) on their OCD symptoms in a clinically meaningful way without exacerbation of bipolar symptoms.

DETAILED DESCRIPTION:
As no systemic data is available regarding the efficacy and safety of selective serotonin reuptake inhibitors (SSRI) in the treatment of OCD+BPD children, it calls for a preliminary open pilot treatment study to explore these issues as a logical first step that could lead to systematic randomized controlled trials in the future. SSRI's are the first line and most commonly used anti-OCD agents. It remains unknown, which of the standard SSRIs is least activating for youth with BPD. Fluoxetine along with fluvoxamine and sertraline are FDA approved for the treatment of OCD in children. Fluoxetine remains the most extensively studied SSRI in children. We will test the safety and efficacy of fluoxetine in children and adolescents with BPD and OCD.

The proposed study includes 1.) the use of a 12-week design to document the response rate and 2.) careful assessment of safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 6 and 17 years of age.
* Participants must have DSM-IV diagnosis of OCD and bipolar (I or II) disorder, displaying current OCD symptoms of at least moderate impairment (CY-BOCS ≥ 15) and for at least 4 weeks prior to participation maintained on steady dose of mood stabilizing medication (lithium, anticonvulsants or atypical antipsychotics) with minimal or mild mood symptoms (YMRS ≤ 15). Period of mood stabilization will be determined by clinician judgment and confirmed by K-SADS-E.
* Subject and his/her legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and his/her legal representative must be considered reliable.
* Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative and the subject must sign an IRB approved informed consent and assent document respectively.
* Subject must be able to participate in mandatory blood draws.
* Subject must be able to swallow pills.
* Subjects with comorbid ADHD, ODD, CD, or other anxiety disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusion Criteria:

* DSM-IV substance dependence (except nicotine or caffeine) within past 3 months.
* History of anti-depressant induced mania or hypomania while also being treated with appropriate dosage(s) of mood stabilizers.
* Pregnant or nursing females.
* Investigator and his/her immediate family, defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Serious, unstable systemic illness.
* History of severe allergies or multiple adverse drug reactions.
* Non-febrile seizures without a clear and resolved etiology.
* Clinically judged to be at serious suicidal risk.
* Other concomitant medication with primary central nervous system activity other than those specified in the Concomitant Medication protocol.
* History of allergic reaction to SSRIs.
* Participants using an MAOI within two weeks prior to receiving study medication.
* Current diagnosis of schizophrenia.
* Uncorrected hypo or hyperthyroidism.
* Active symptoms of anorexia or bulimia nervosa
* Non-response of OCD symptoms to fluoxetine as defined by being on therapeutic dose of fluoxetine for at least 10 weeks.
* Current treatment with antidepressant medication.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2005-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluoxetine
Started | 13
Completed | 7
Not Completed | 6
Not completed — Non-compliance | 1
Not completed — Adverse Event | 3
Not completed — Found ineligible | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fluoxetine
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.46 (3.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: This sale measures impairment on 5 items relating to Obsessions from 0 (none) to 4 (extreme) and 5 item relating to Compulsions from 0 (none) to 4 (extreme). These scores are totaled for a range of 0 (least impaired) to 40 (most impaired).
Time Frame: weekly
Population: 2 participants were not included in final analysis - 1 terminated at 1 week due to non-compliance with taking study medication. 1 found ineligible prior to beginning treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 11
Units on a scale | 14.18 (9.98)

2. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: This scale measures mania symptoms in children and adolescents using 11 items rated from 0 (least severe) to 4 (most severe), although 4 items are rated from 0-8. The minimum (least severe) possible score is 0, and the maximum (most severe) possible score is 60.
Time Frame: weekly
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoxetine
Number analyzed (Participants) | 11
Units on a scale | 13 (12.54)

ADVERSE EVENTS:
Arm/Group | Fluoxetine
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=11)
bilateral medial thigh skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
blurred vision (distance) (Eye disorders) | 1 (1)
chest uneasiness (General disorders) | 1 (1)
decreased appetite (General disorders) | 1 (1)
dizziness (Ear and labyrinth disorders) | 2 (3)
drooling (General disorders) | 1 (3)
eczema rash (Skin and subcutaneous tissue disorders) | 1 (1)
frequent urination (Renal and urinary disorders) | 1 (1)
headache (General disorders) | 2 (4)
hurt cheek playing soccer (Injury, poisoning and procedural complications) | 1 (1)
increased appetite (General disorders) | 3 (8)
irritable (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
nose bleed (General disorders) | 1 (1)
runny nose (General disorders) | 1 (1)
sleep disturbance (General disorders) | 1 (1)
tiredness (General disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 1 (1)
worsening of manic symptoms (Psychiatric disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes